CLINICAL TRIAL: NCT06023511
Title: Safety and Efficacy of the MyokinE100 (CL-EMS Alpha) Device in Inducing Visible Muscle Contraction in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Discovery Labs (Industry)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); University of Texas at Austin (Other); Ascension Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY00004235
Record Dates: First submitted 2023-08-23; First posted 2023-09-05 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: ICU Acquired Weakness
Keywords: Muscle weakness; Critical care myopathy; Electrical muscle stimulation; Electromagnetic interference; ICU monitoring
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Intervention group (Experimental): Volunteers will receive electrical muscle stimulation.
  Interventions: Device: Electrical muscle stimulation

INTERVENTIONS:
Device: Electrical muscle stimulation — While study subjects are connected to standard ICU monitors, electrical muscle stimulation will be applied at the level of the quadriceps muscle to induce palpable or visible muscle contraction. (No control group or sham procedure in this study).
  Other Names: MyokinE100 (CL-EMS alpha)

SUMMARY:
Every patient admitted to the Intensive Care Unit (ICU) is at risk of developing "Intensive Care Unit Acquired Weakness" (ICUAW). ICUAW is associated with increased rate of mortality, prolonged duration of mechanical ventilation, ICU and hospital stay, rehabilitation time, and reduced quality of life. Currently, there is no effective treatment for ICUAW.

Health Discovery Labs is conducting a research study to evaluate the safety of using an innovative experimental medical device in ICU settings that could mitigate ICUAW.

This study is meant to demonstrate whether this new device interferes with standard ICU monitors.

DETAILED DESCRIPTION:
Every patient admitted to the ICU is at risk of developing ICU Acquired Weakness (ICUAW). ICUAW begins within the first couple hours of hospitalization with approximately 11% of muscle strength is lost per day. Further, 2.4 million patients per year in the US develop an advanced form of ICUAW which is associated with increased rate of mortality, prolonged duration of mechanical ventilation, ICU and hospital stay, rehabilitation time, and reduced quality of life. To mitigate ICUAW, early mobility is the lone strategy readily available to clinicians to thwart ICUAW. Early mobility programs require patient's cooperation and numerous ICU staff safely implement the intervention. Thus, uncooperative patients are excluded from mobility efforts. Clearly, interventions that can be implemented with most any ICU patient are urgently needed. Electrical muscle stimulation (EMS) is uniquely capable of addressing this need by contracting muscles using skin-surface electrodes and electrical pulses. Clinical data assessing the feasibility, safety, and efficacy of such intervention is promising. However, technical limitations such as lack of electric safety in commercially available devices, and the need for a skilled operator to install, setup, and monitor the treatment session render the application of electrical muscle stimulation as a tool for early rehabilitation in the ICU complex and expensive. To solve this problem, Health Discovery Labs is developing an easy-to-use closed loop electrical muscle stimulation system (CL-EMS) with improved electric safety. The objective of this interventional, open label single group feasibility study is to assess whether the MyokinE100 (CL-EMS alpha) device developed by Health Discovery Labs will interfere with cardiac monitoring devices commonly used in ICU settings while inducing muscle contraction or twitching.

In Simulation Lab ICU setting, at the Ascension Texas Clinical Education Center (CEC), healthy volunteers will be placed in supine position on an electrically powered ICU bed, connected to the cardiac monitor system, and to an external defibrillator in monitor mode. A pair of garments containing off-the-shelf (OTS) electrodes will be wrapped around the thigh area (both right and left lower limb) and connected to the MyokinE100 (CL-EMS alpha) device developed by Health Discovery Labs. Volunteers will receive electrical muscle stimulation of contralateral muscle groups for a total of 25 minutes. Before and during the electrical muscle stimulation process, data related to the ECG patterns will be collected from the ECG monitoring system, and the external defibrillator. Data related to the applied electrical pulse characteristics will be collected from the device. Muscle response to electrical stimulation will be objectively graded by the research team based on a scale for rating the quality of muscle contractions. Comfort level will be graded by the volunteer using the Numeric Rating Scale (NRS).

Success will be judged based on the following criteria: (1) the use of the MyokinE100 (CL-EMS alpha) device does not induce ECG noise of more than 0.1mV in amplitude in at least 70% of the healthy volunteers; (2) does not introduce signals suggestive of cardiac dysrhythmias (VF/VT/AF/PVC/PAC) in at least 70% of the healthy volunteers; and (3) induces visible muscle contraction at the level of the quadriceps muscle group in at least 70% of the healthy volunteers.

ELIGIBILITY:
Inclusion:

* Male or female
* Age 18 to 65
* Healthy volunteers with no significant past medical history

Exclusion:

* History of heart disease
* Family history of sudden cardiac death
* History of neurological or neuromuscular diseases, or genetic muscular disorders
* History of deep vein thrombosis
* Presence of implantable devices
* Recent hospitalization within the last 3-months (surgical or medical)
* Pregnancy
* Allergy to latex
* Allergy to carbon-based electrodes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
Interference with cardiac monitoring devices: detection of ECG noise of more than 0.1mV in amplitude or ECG changes suggestive of cardiac dysrhythmias | During the 25 minutes that the EMS is applied to each test subject.
  During electrical muscle stimulation using the MyokinE100 (CL-EMS alpha) device at the level of the quadriceps muscle, volunteers will be connected to cardiac monitoring device. ECG will be monitored for the detection of electric interference or the detection of noise suggestive of dysrhythmias.
  Success will be based on the following criteria: (1) intervention does not induce noise of more than 0.1mV in amplitude; and (2) does not introduce signal suggestive of cardiac dysrhythmias (VT/VF/AF/PVC/PAC)

SECONDARY OUTCOMES:
Grading of muscle contraction to electrical stimulation using the scale for rating the quality of muscle contractions. | During the 25 minutes that the EMS is applied to each test subject.
  Evaluate the type of muscle contraction generated by the device in healthy volunteers using the scale of muscle contractions published by Gosselink et al. [PMID 25108833].
  Type 1 = No palpable or visible contraction; Type 2 = Just palpable but no visible contraction; Type 3 = Just palpable and just visible contraction; Type 4 = Palpable and visible contraction (partial muscle bulk); Type 5 = Palpable and visible contraction (full muscle bulk).

CONTACTS AND LOCATIONS:
Overall Officials: Oussama Hassan, MD, Study Director — Health Discovery Labs LLC; Paul Harford, MD, Principal Investigator — University of Texas at Austin
Locations (1):
- Ascension Texas Clinical Education Center (CEC), Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ICU-acquired weakness and recovery from critical illness — https://pubmed.ncbi.nlm.nih.gov/24758618/
- See also: Feasibility of neuromuscular electrical stimulation in critically ill patients — https://pubmed.ncbi.nlm.nih.gov/25108833/